CLINICAL TRIAL: NCT02062476
Title: EPIGENETIC EFFECTS ELICITED BY LACTOBACILLUS GG IN CHILDREN WITH COW'S MILK ALLERGY: A POSSIBLE EFFECT OF ATOPIC MARCH
Brief Title: Epigenetic Effects Elicited By Lactobacillus GG In Children With Cow's Milk Allergy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/14
Record Dates: First submitted 2014-02-06; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

ARMS (2):
- Treatment with Lactobacillus GG (Experimental): extensively hydrolyzed casein formula containing LGG
  Interventions: Dietary Supplement: Lactobacillus GG
- Children at diagnosis (No Intervention)

INTERVENTIONS:
Dietary Supplement: Lactobacillus GG
  Arms: Treatment with Lactobacillus GG

SUMMARY:
Lactobacillus GG (LGG) is able to exert long lasting effects in children with atopic disorders. We have shown that Nutramigen LGG accelerates tolerance acquisition in infants with cow's milk allergy (CMA). The mechanisms of these effects are still largely undefined. The effect of LGG could be related at least in part by the immunoregulatory role played by LGG. This probiotic can balance the generation of cytokines possibly involved in IgE- or non-IgE-mediated CMA (i.e., IL-4, IL-5, IL-10, IFN-γ , TGF-beta, and TNF-alfa), which can contribute to modulation of inﬂammatory processes. We have demonstrated that children with IgE-mediated CMA produce significantly higher level of IL-4 and IL-13 in response to cow's milk protein, and that tolerance is associated with a marked reduction of IL-13 production and a concomitant increased frequency of IFN-γ releasing cells.

Epigenetics studies the heritable (and potentially reversible) changes of the genome inherited from one cell generation to the next which alter gene expression but do not involve changes in primary DNA sequences, highlighting the complexity of the inter-relationship between genetics and nutrition. There are three distinct, but closely interacting, epigenetic mechanisms (histone acetylation, DNA methylation, and non-coding microRNAs) that are responsible for modifying the expression of critical genes associated with physiologic and pathologic processes. The profile of epigenetic modifications associated with Th lineage commitment, coupled with the sensitivity of the early developmental period, has led to speculation that factors that disrupt these pathways may increase the risk of allergic diseases. Specifically, effects on DNA methylation and endogenous histone deacetylase inhibitors acting on specific pathways (Th1 and T regulatory cell differentiation) may favour Th2-associated allergic differentiation. MicroRNAs are another structural components of an epigenetic mechanism of post-transcriptional regulation of messenger RNA translation. It has been recently identified a specific Th2-associated miRNA (miR-21) that is critical for the regulation of Th cell polarization.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 months-4 years with cow's milk allergy

Exclusion Criteria:

* age higher than 4 years,
* concomitant chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal tract,
* suspected eosinophilic esophagitis or eosinophilic enterocolitis,
* suspected food-protein-induced enterocolitis syndrome,
* suspected cow's milk protein-induced anaphylaxis.

Ages: 4 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 6 months in tolerance acquisition and epigenetic effects in rtwenty children with cow's milk allergy | Baseline, at least after 6 months of therapy
  The investigators will evaluate in children with CMA if the effect of Lactobacillus GG on tolerance acquisition is mediated at least in part by an epigenetic mechanism.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy